CLINICAL TRIAL: NCT01476540
Title: Deep Brain Stimulation for the Treatment of Refractory Anorexia Nervosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Andres M. Lozano, Neurosurgeon, Professor of Surgery, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-0991-A
Record Dates: First submitted 2011-11-15; First posted 2011-11-22 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Deep Brain Stimulation (Experimental): Deep Brain Stimulation
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — Deep Brain Stimulation (DBS) is a neurosurgical procedure involving the implantation of deep brain electrodes, connected via a subcutaneous extension wire, to an implantable pulse generator (IPG, or 'battery') that is implanted below the collarbone.

SUMMARY:
Anorexia Nervosa (AN) is a challenging, chronic, refractory illness with the highest mortality rate of any psychiatric condition. Advances in the neuroimaging, genetics and neurobiology of AN has led to a greater understanding of its underlying pathophysiology, although few significant advances in treatment have been made in the last half-century. The central features of AN, which include an intense fear of gaining weight, a refusal to maintain a normal weight, as well as significant anxiety, anhedonia and dysphoria surrounding food, have been linked to dysfunction in key brain structures and circuits. Deep Brain Stimulation (DBS) is a neurosurgical procedure that involves the insertion of electrodes into structures believed to drive pathological behavior. The procedure is approved for the management of movement disorders, such as Parkinson's Disease, and has shown promising early results in the management of some psychiatric conditions, such as Major Depression. The purpose of this study is to explore the safety and initial efficacy of DBS, in patients with treatment resistant AN.

DETAILED DESCRIPTION:
Anorexia nervosa is a chronic, and debilitating psychiatric disorder associated with the highest mortality rate of any psychiatric condition. Despite advances in neuroimaging, genetics, pharmacology and psychosocial interventions in the last half century, little progress have been made in altering the natural history of the condition or its outcomes. It has further become increasingly accepted that the thoughts and behaviors at the root of AN derive from dysfunctional neuroanatomic circuits, whose activity and deviations can be detected with sophisticated neuroimaging techniques. Much progress has also been made in mapping the psychology of the illness to underlying neuroanatomic and neurophysiologic processes that drive and maintain these behaviors, even in the face of severe starvation and impending death. Dysfunctional reward processing, compulsive hyperactivity, chronic anxiety and depression, all suggest that AN shares much in common with other conditions, such as OCD, for which surgical therapy has been tried, and met with success.

Deep Brain Stimulation is a neurosurgical tool that has been widely used for over twenty years. Most of the experience with DBS comes from the movement disorder literature where significant success has been had with the management of disabling Parkinson's disease (PD) and dystonia. The most experience so far has been in Parkinson's disease where well over 50,000 patients globally have received the operation. DBS is believed to work by using small amounts of electricity to disrupt the activity of brain structures that produce troublesome symptoms. DBS has also been used in psychiatric patients, both as part of treatment and research, in cases of Obsessive-Compulsive Disorder (OCD), and research, in cases of Depression. Current research suggests that there are similarities between Anorexia Nervosa and conditions such as OCD and depression. Given that DBS has shown promise in the treatment of those conditions, this trial was designed to see if it could be an effective therapy for Anorexia Nervosa as well.

This study would be the first exploration of a surgical therapy for refractory AN. The rationale stems from clear and robust evidence pointing at a dysfunctional cortical-subcortical loop driving abnormal behavior, with several important nodes in the loop being particularly important, and recurring, players. The subgenual cingulate plays a role in affective decision making, reward processing, as well as subsequent anxiety and dysphoric mood.

There are currently no brain based, targeted therapies for AN. The scientific significance of this study will be:

i) The first clinical trial exploring deep brain stimulation in an eating disorder population

ii) The first demonstration of the influence of deep brain stimulation on dysfunctional reward processing with co-morbid anxiety/dysphoria

iii) The first 'brain-based' treatment for any eating disorder

ELIGIBILITY:
Inclusion Criteria:

* Female or Male patients between age 20-60
* Diagnosis of Anorexia Nervosa, restricting or binge-purging subtype as defined by the Diagnostic and Statistical Manual (DSM-IVR)
* Chronicity and/or Treatment Resistance as demonstrated by some or all of:

  1. A pattern of three year's duration of relentless unresponsiveness to repeated voluntary hospitalizations, characterized by failure to complete treatment of immediate weight relapse following treatment;
  2. pattern of increasing medical instability accompanied by refusal to participate in/lack of responsiveness to intensive expert treatment and increasing medical acuity, lasting at least two years and involving at least two episodes of involuntary feeding;
  3. A pattern of chronic stable AN lasting at least 10 years
* Able to comply with all testing, follow-ups and study appointments and protocols

Exclusion Criteria:

* Any past or current evidence of psychosis
* Active neurologic disease such as epilepsy
* Alcohol or substance dependence or abuse in the last 6 months, excluding caffeine and nicotine
* Any contraindication to Magnetic Resonance Imaging (MRI) or Positron Emission Tomography (PET) scanning
* Likely to relocate or move during the study's one year duration
* BMI less than 13
* Presence of cardiac arrhythmias, or other cardiac, respiratory, renal or endocrine conditions as a result of AN or not, that will result in significant risk from a surgical procedure.
* Pregnancy

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2011-07; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Eating Disorder Related Preoccupations and Rituals | Change from baseline in Eating Disorder Related Preoccupations and Rituals scores at 3 months, 6 months and 12 months
  Eating Disorder Related Preoccupations and Rituals scores

SECONDARY OUTCOMES:
Depression | Change from baseline in depression scores at 3 months, 6 months and 12 months
  Hamilton Depression Rating Scale (HAMD), Beck Depression Inventory (BDI)
Anxiety | Change from baseline in anxiety scores at 3 months, 6 months and 12 months
  Beck Anxiety Inventory (BAI)
Quality of Life questionnaire score through change from baseline compared to post-implant visit | Change from baseline in Quality of Life scores at 3 months, 6 months and 12 months
  Health Survey Short Form (SF36), Quality of Life Scale

CONTACTS AND LOCATIONS:
Overall Officials: Andres M Lozano, MD, PhD, Principal Investigator — University Health Network, Toronto; Blake Woodside, MD, Principal Investigator — Toronto General Hospital
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Lipsman N, Lam E, Volpini M, Sutandar K, Twose R, Giacobbe P, Sodums DJ, Smith GS, Woodside DB, Lozano AM. Deep brain stimulation of the subcallosal cingulate for treatment-refractory anorexia nervosa: 1 year follow-up of an open-label trial. Lancet Psychiatry. 2017 Apr;4(4):285-294. doi: 10.1016/S2215-0366(17)30076-7. Epub 2017 Feb 24. PMID 28238701
- [Derived] Lipsman N, Woodside DB, Giacobbe P, Hamani C, Carter JC, Norwood SJ, Sutandar K, Staab R, Elias G, Lyman CH, Smith GS, Lozano AM. Subcallosal cingulate deep brain stimulation for treatment-refractory anorexia nervosa: a phase 1 pilot trial. Lancet. 2013 Apr 20;381(9875):1361-1370. doi: 10.1016/S0140-6736(12)62188-6. Epub 2013 Mar 7. PMID 23473846